CLINICAL TRIAL: NCT05489809
Title: Endotracheal Extubation With Suctioning Versus Positive Pressure in Children After General Anaesthesia. A Randomised Control Trial.
Brief Title: Endotracheal Extubation With Suctioning Versus Positive Pressure in Children After General Anaesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Navy Station Shifa Hospital (Other)
Responsible Party: Principal Investigator, Kenan Anwar Khan, Graded Anaesthetist, Principal Investigator, Pakistan Navy Station Shifa Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERC/2022/ANS/2
Record Dates: First submitted 2022-07-26; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Endotracheal Extubation
MeSH Terms: interventions — Airway Extubation; Suction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotracheal extubation with suctioning (Experimental): Suctioning is applied to the endotracheal tube while removing it.
  Interventions: Procedure: Endotracheal extubation with suctioning
- Endotracheal extubation with positive pressure (Experimental): Positive pressure is applied to the endotracheal tube while removing it.
  Interventions: Procedure: Endotracheal extubation with positive pressure

INTERVENTIONS:
Procedure: Endotracheal extubation with suctioning — General anestheisa is maintained with an endotracheal tube. At the end of anesthesia, the endotracheal tube is removed by applying suctioning.
  Arms: Endotracheal extubation with suctioning
Procedure: Endotracheal extubation with positive pressure — General anesthesia is maintained with an endotracheal tube. At the end of anesthesia, the endotracheal tube is removed by applying positive pressure.
  Arms: Endotracheal extubation with positive pressure

SUMMARY:
Comparing extubation of endotracheal tube in children after general anaesthesia by applying suctioning to the endotracheal tube versus applying positive pressure to the endotracheal tube.

DETAILED DESCRIPTION:
Extubation after general anaesthesia involves removal of the endotracheal tube. This is done by either applying suctioning or applying positive pressure to the endotracheal tube. My study aims at identifying which technique is superior to the other.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II patients
* either sex
* consent given

Exclusion Criteria:

* not meeting the inclusion criteria

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Endotracheal extubation | 3 months
  The intervention will try to identify which technique is better to extubate the patient after general anesthesia.
  In literature/anesthesia practice there is no scale, parameter or questionnaire to indicate extubation. However the aim is universally accepted that is to extubate the patient when he/she is hemodynamically stable and able to maintain a patent airway and oxygen saturation while spontaneously breathing and awake.
  In my trial, half the number of participants will be extubated by applying suctioning to the endotracheal tube and the remaining will be extubated by applying positive pressure to the endotracheal tube at the end of general anesthesia.
  Patients heart rate, blood pressure, oxygen saturation, the need for clearing secretions from the airway, and the need for supplemental oxygen at the time of extubation and 3 minutes after extubation will be compared to identify which technique is better in terms of patients airway management.

SECONDARY OUTCOMES:
Pulse | 3 months
  Heart rate in beats per minute
Oxygen saturation | 3 months
  Oxygen saturation in percentage
Blood pressure | 3 months
  Blood pressure in millimetre of mercury
Supplemental oxygen | 3 months
  Supplemental oxygen in liters per min
Airway suctioning | 3 months
  Number of times suctioning required to clear airway secretions

CONTACTS AND LOCATIONS:
Overall Officials: Kenan Khan, Principal Investigator — Pakistan Navy Station Shifa Hospital
Locations (1):
- PNS Shifa Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No